CLINICAL TRIAL: NCT02736643
Title: Retrospective Epidemiological Study of Lung Cancer With Low-dose Multislice Computed Tomography (LDCT) - a Screening Program
Brief Title: Retrospective Epidemiological Study of Lung Cancer With Low-dose Multislice Computed Tomography
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201601052RINB
Record Dates: First submitted 2016-04-10; First posted 2016-04-13 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: LDCT, screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
Lung cancer is one of the leading causes of cancer-related death in Taiwan. Early diagnosis of lung cancer may improve cancer survival. Low-dose computed tomography (LDCT) was thought to be the best screening tool for lung cancer. However, there is growing concerns about radiation exposure, high cost, and high rate of false-positive screening result. Epidemiology data for LDCT screening in Taiwan is lacking.

National Taiwan University Hospital Chu-Tung Branch (NTUHCT) initiated the lung cancer screening by LDCT since June 2015. Many people can get the LDCT screening with affordable price with the subsidy from enterprise donation. The purpose of this study is establishing local epidemiological result via telephone follow-up and patients' medical records retrospectively.

DETAILED DESCRIPTION:
Lung cancer is one of the leading causes of cancer-related death in Taiwan. Early diagnosis of lung cancer may improve cancer survival. Low-dose computed tomography (LDCT) was thought to be the best screening tool for lung cancer. However, there is growing concerns about radiation exposure, high cost, and high rate of false-positive screening result. Epidemiology data for LDCT screening in Taiwan is lacking.

National Taiwan University Hospital Chu-Tung Branch (NTUHCT) initiated the lung cancer screening by LDCT since June 2015. Many people can get the LDCT screening with affordable price with the subsidy from enterprise donation. The purpose of this study is establishing local epidemiological result via telephone follow-up and patients' medical records retrospectively.

Aim: To establish the local epidemiological data for lung pathology, emphysema, bronchiectasis and other lung disease.

Methods: Since June 2015, more than 6000 LDCT were done at the NTUHCT. Roughly 6 months after the test telephone follow-ups about patient satisfactions, self-awareness of CT results, medical consultations and other related behaviors, and willingness of coming back for another test were routinely done. Retrospective secondary data analysis will be performed on the telephone follow-up results to establish local epidemiology data on lung pathology as well as information on screening accuracy of LDCT. Customers are also queried about willingness to provide their medical records, and linkage to National Health Insurance Database with informed consents to provide more advanced information on their long-term outcomes.

Keywords: Lung cancer, Low dose computed tomography, screening.

ELIGIBILITY:
Inclusion Criteria:

* self pay the LDCT in National Taiwan University Hospital Chu-Tung Branch

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: self pay the LDCT in National Taiwan University Hospital Chu-Tung Branch
Sampling Method: Probability Sample
Enrollment: 1334 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12-28 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Abnormal lung finding detection rate | one month
  Abnormal lung finding detection rate calculated as (patients with abnormal finding from LDCT / total enrollments).

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital Chu-Tung Branch

IPD SHARING:
Plan to Share IPD: No